CLINICAL TRIAL: NCT05458999
Title: Decreasing Patient Anxiety During Percutaneous Revascularization of Chronic Total Coronary Occlusions Using Virtual Reality Glasses.
Brief Title: Decreasing Patient Anxiety During Revascularization of Chronic Total Coronary Occlusions Using Virtual Reality Glasses.
Acronym: ReViCTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Agustín Fernández, Interventional Cardiologist, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/031
Record Dates: First submitted 2022-06-29; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Chronic Total Occlusion; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, prospective, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality headset (Experimental): Virtual reality headset during percutaneous coronary intervention
  Interventions: Other: Virtual reality headset during percutaneous coronary intervention
- Control (No Intervention): Routine clinical practice

INTERVENTIONS:
Other: Virtual reality headset during percutaneous coronary intervention — Virtual reality glasses during percutaneous coronary intervention
  Arms: Virtual reality headset

SUMMARY:
Percutaneous coronary angioplasty on chronic total occlusions is a complex procedure. The possibility of performing these procedures without anesthesia and sedation avoids the risks associated with anesthesia and sedation, but, on the contrary, subjects the patient to pain and anxiety during the procedure.

Virtual reality (VR) has been successfully used in several clinical settings to reduce intra-procedural anxiety.

The aim of this clinical trial is to determine whether the use of a VR system in PCI procedures on CTO decreases the level of anxiety and pain during the procedure.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) on chronic total occlusions (CTO) represents one of the greatest challenges in interventional cardiology, due to the complexity of these procedures and the increased risk of complications. In recent decades, advances in techniques and devices have made it possible to obtain better results while reducing the associated complications.

The possibility of performing these procedures without anesthesia or sedation avoids the risks derived from these, but, on the contrary, subjects the patient to pain and anxiety during the procedure. Several factors influence patient anxiety: long duration of procedures, patient immobility (especially in biradial access), monotonous and hostile environment (operating rooms or catheterization rooms). Anxiety and pain are treated by pretreatment with oral benzodiazepines supplemented by opioids or intravenous benzodiazepines on demand during the procedure, assuming the possible complications derived from this treatment.

Virtual reality (VR) has been used successfully in several clinical settings to reduce intra-procedural anxiety. A reduction in anxiety and pain has been demonstrated even in elderly patients undergoing percutaneous aortic valve replacement. Its use does not require technical expertise or experience in the use of digital devices and does not increase the sensation of dizziness or nausea.

The aim of this study is to determine whether the use of a VR system in PCI procedures over CTO decreases the level of anxiety and pain during the procedure.

Method

Design Randomized, single-center, prospective, open-label study. Each patient will be assigned by simple randomization (in a 1:1 ratio) to intervention group (use of VR goggles during the CTO procedure) or control group (usual practice). Randomization will be performed once the patient is in the catheterization laboratory.

Population After signing the informed consent form, all patients undergoing programmed PCI on CTO performed at the Hospital Clínico Universitario de Valencia from 01/12/2021 will be consecutively included until the calculated sample size is completed. Patients with visual deficits, dementia, language barrier or any other situation that prevented the use of VR glasses will be excluded.

Objectives The primary objective will be the maximum level of anxiety perceived by the patient measured by a visual analog scale (VASa) (1-10) and determined at the end of the procedure. Secondary objectives will be the level of pain perceived by the patient using a visual analog scale (VASd), the need for intraprocedural anxiolytic pharmacological treatment, the dose of drug administered and the degree of satisfaction with the VR goggles.

Both VASa and VASd will be collected by a specialist nurse just after the end of the procedure, and before leaving the room by means of a specific questionnaire.

Sample size calculation. A sample size of 58 patients, 29 in each group, was calculated to detect a difference equal to or greater than 2 points assuming an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast. The common standard deviation for VASa was assumed to be 2.7.

Data management. Variables will be collected in an electronic data collection notebook for each patient 1. Demographics (age, sex), 2. History: Cardiovascular risk factors (arterial hypertension, hypercholesterolemia, diabetes mellitus), cardiological history (acute myocardial infarction, ischemic heart disease, percutaneous coronary intervention, coronary revascularization surgery, heart failure, stroke), usual pharmacological treatment (antiplatelet agents, beta-blockers, nitrates, calcium antagonists, ranolazine, statins, diuretics, antidiabetics, antidepressants, benzodiazepines, hypnotics), 3. Preprocedure: Seattle Angina Questionnaire (SAQ), dyspnea (New York Heart Association functional class -NYHA), indication for revascularization (persistent angina despite optimal medical treatment, silent ischemia), ischemia screening test (MRI, stress echocardiogram), previous analytical (creatinine, hemoglobin, amino-terminal pro-B-type natriuretic peptide -NTproBNP), ejection fraction, number of previous CTO revascularization attempts, familiarity with new technologies, 4. Periprocedural: accesses (one or two femoral accesses, biradial, radial-femoral), total duration of procedure, total escopia time, radiological dose (dose-area product, Kerma in air), VASa (measured before room entry and peak level during the procedure), administered dose of morphine chloride, midazolam or other anxiolytics, maximum level of chest pain during the procedure (visual scale), nausea, dizziness, overall satisfaction with the procedure (visual analog scale) and overall satisfaction with the use of VR headset.

Intervention A commercial Oculus Quest 2 virtual reality headset system (Facebook Technologies, LLC, California (USA) will be used. Using the Netflix video streaming system application (Netflix Inc. California (USA) the documentary series "Our Planet" (Silverback Films, UK) will be screened for all patients, starting with chapter 1 and sequentially and automatically playing the following chapters. Before the procedure, the patient will be informed of the operation of the VR goggle system and possible side effects (nausea or dizziness) as well as the possibility of removing it at any time. Before starting the arterial puncture, the VR headset system will be put on and checked for proper functioning. It will be removed prior to removal of the arterial introducers, when the patient expresses a desire to remove it or if serious complications occur. During the procedure, the patient's general condition will be checked every 30 minutes.

In both groups, the administration of anxiolytic drugs (morphine chloride or midazolam in 1 mg boluses) will be at the discretion of the main operator and according to the degree of anxiety perceived. The rest of the actions for the management of pre- and peri-procedure anxiety will be identical in both groups.

Statistical analysis Quantitative variables will be expressed as mean ± standard deviation when they follow a normal distribution and as median [interquartile range] when they do not. Quantitative variables will be expressed as percentages (absolute value). The Fisher or Chi-square test will be used to compare qualitative variables and the Student t test (or Mann-Whitney U test, in the case of not following a normal distribution) for quantitative variables.

All statistical tests will be bilateral and considered significant at p<0.05. Statistical analyses will be performed with R Core Team (2020) software (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Chronic total oclussion scheduled percutaneous coronary intervention.

Exclusion Criteria:

* Less than 18 years old.
* Visual deficits
* Dementia
* Language barrier
* Any other situation that would prevent the use of VR goggles.
* Inability or refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Intraprocedure
  Maximum level of anxiety perceived by the patient measured by a visual analog scale (VASa) (1-10) and determined at the end of the procedure.

SECONDARY OUTCOMES:
Pain level | Intraprocedure
  Maximum pain level perceived by the patient measured by a visual analog scale (VASa) (1-10) and determined at the end of the procedure.
Need of anxiolytic treatment | Intraprocedure
  Need of anxiolytic farmacological treatment (opioids or benzodiazepines) during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No